CLINICAL TRIAL: NCT06305572
Title: Diagnostic Accuracy of Quantitative Flow Ratio for Hemodynamic Assessment of Coronary Artery Stenosis: Prospective Observational Study
Brief Title: Diagnostic Accuracy of Quantitative Flow Ratio
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University Ilsan Paik Hospital (Other); Keimyung University Dongsan Medical Center (Other); Ulsan Medical Center (Other); Sejong General Hospital (Other); Chosun University Hospital (Other); Severance Hospital (Other); Ulsan University Hospital (Other); Uijeongbu Eulji Medical Center (Unknown)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: H-1903-013-1014
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QFR group: Patients suspected with coronary artery disease undergoing diagnostic coronary angiography with an indication for to perform invasive FFR
  Interventions: Diagnostic Test: QFR

INTERVENTIONS:
Diagnostic Test: QFR — Patients suspected with CAD undergoing diagnostic coronary angiography with an indication for to perform invasive FFR were included. QFR was analyzed in an independent core laboratory (Uijeongbu Eulji Medical Center) using the software package QAngio XA 3D 2.1 (Medis Medical Imaging Systems, Leiden, the Netherlands).

SUMMARY:
The aim of this study was to investigate the accuracy of quantitative flow ratio (QFR) for predicting fractional flow reserve (FFR) ≤0.80 in an independent core laboratory.

DETAILED DESCRIPTION:
FFR is an invasive physiological index used to define coronary stenosis that causes ischemia. Several studies have suggested that FFR-based percutaneous coronary intervention (PCI) can reduce adverse clinical outcomes compared to angiography-guided PCI. Although FFR is highly recommended in current guidelines, it is underused in real-world practice. QFR is a method for evaluating fractional flow reserve FFR without the use of an invasive coronary pressure wire or pharmacological hyperemic agent.

The aims of this study were:

1. To investigate diagnostic accuracy of angiography-based QFR for hemodynamic assessment of coronary artery stenosis compared to pressure wire-based FFR.
2. To compare the diagnostic performance of QFR versus % diameter stenosis (DS) in identifying physiologically significant coronary artery disease (CAD) using FFR as the reference standard.
3. To identify factors affecting QFR accuracy.
4. To compare the coronary CT data with QFR.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected with CAD undergoing diagnostic coronary angiography with an indication for to perform invasive FFR

Exclusion Criteria:

* Suboptimal angiographic image quality for QFR analysis
* Primary myocardial or valvular disease
* Left ventricular ejection fraction ≤40%
* Patients with cardiogenic shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected with CAD undergoing diagnostic coronary angiography with an indication for to perform invasive FFR were included. Clinical exclusion criteria included cardiogenic shock, reduced ejection fraction (EF ≤40%), or suboptimal angiographic image quality for QFR analysis.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of QFR | through study completion, an average of 1 year
  Diagnostic accuracy of QFR (≤0.80 or >0.80) to determine hemodynamically significant coronary stenosis using invasive FFR (≤0.80 or >0.80) as a reference standard

SECONDARY OUTCOMES:
Sensitivity of QFR | through study completion, an average of 1 year
  Sensitivity of contrast QFR to predict FFR lower than 0.8
Specificity of QFR | through study completion, an average of 1 year
  Specificity of contrast QFR to predict FFR lower than 0.8
Correlation | through study completion, an average of 1 year
  Correlation between QFR and FFR

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The sharing plan will be decided by the study committee.

REFERENCES:
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] van Nunen LX, Zimmermann FM, Tonino PA, Barbato E, Baumbach A, Engstrom T, Klauss V, MacCarthy PA, Manoharan G, Oldroyd KG, Ver Lee PN, Van't Veer M, Fearon WF, De Bruyne B, Pijls NH; FAME Study Investigators. Fractional flow reserve versus angiography for guidance of PCI in patients with multivessel coronary artery disease (FAME): 5-year follow-up of a randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1853-60. doi: 10.1016/S0140-6736(15)00057-4. Epub 2015 Aug 30. PMID 26333474
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Pijls NH, Fearon WF, Tonino PA, Siebert U, Ikeno F, Bornschein B, van't Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, De Bruyne B; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention in patients with multivessel coronary artery disease: 2-year follow-up of the FAME (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation) study. J Am Coll Cardiol. 2010 Jul 13;56(3):177-84. doi: 10.1016/j.jacc.2010.04.012. Epub 2010 May 28. PMID 20537493
- [Background] Gotberg M, Cook CM, Sen S, Nijjer S, Escaned J, Davies JE. The Evolving Future of Instantaneous Wave-Free Ratio and Fractional Flow Reserve. J Am Coll Cardiol. 2017 Sep 12;70(11):1379-1402. doi: 10.1016/j.jacc.2017.07.770. PMID 28882237
- [Background] Tu S, Westra J, Yang J, von Birgelen C, Ferrara A, Pellicano M, Nef H, Tebaldi M, Murasato Y, Lansky A, Barbato E, van der Heijden LC, Reiber JHC, Holm NR, Wijns W; FAVOR Pilot Trial Study Group. Diagnostic Accuracy of Fast Computational Approaches to Derive Fractional Flow Reserve From Diagnostic Coronary Angiography: The International Multicenter FAVOR Pilot Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2024-2035. doi: 10.1016/j.jcin.2016.07.013. PMID 27712739
- [Background] Westra J, Andersen BK, Campo G, Matsuo H, Koltowski L, Eftekhari A, Liu T, Di Serafino L, Di Girolamo D, Escaned J, Nef H, Naber C, Barbierato M, Tu S, Neghabat O, Madsen M, Tebaldi M, Tanigaki T, Kochman J, Somi S, Esposito G, Mercone G, Mejia-Renteria H, Ronco F, Botker HE, Wijns W, Christiansen EH, Holm NR. Diagnostic Performance of In-Procedure Angiography-Derived Quantitative Flow Reserve Compared to Pressure-Derived Fractional Flow Reserve: The FAVOR II Europe-Japan Study. J Am Heart Assoc. 2018 Jul 6;7(14):e009603. doi: 10.1161/JAHA.118.009603. PMID 29980523
- [Background] Xu B, Tu S, Qiao S, Qu X, Chen Y, Yang J, Guo L, Sun Z, Li Z, Tian F, Fang W, Chen J, Li W, Guan C, Holm NR, Wijns W, Hu S. Diagnostic Accuracy of Angiography-Based Quantitative Flow Ratio Measurements for Online Assessment of Coronary Stenosis. J Am Coll Cardiol. 2017 Dec 26;70(25):3077-3087. doi: 10.1016/j.jacc.2017.10.035. Epub 2017 Oct 31. PMID 29101020
- [Background] Xu B, Tu S, Song L, Jin Z, Yu B, Fu G, Zhou Y, Wang J, Chen Y, Pu J, Chen L, Qu X, Yang J, Liu X, Guo L, Shen C, Zhang Y, Zhang Q, Pan H, Fu X, Liu J, Zhao Y, Escaned J, Wang Y, Fearon WF, Dou K, Kirtane AJ, Wu Y, Serruys PW, Yang W, Wijns W, Guan C, Leon MB, Qiao S, Stone GW; FAVOR III China study group. Angiographic quantitative flow ratio-guided coronary intervention (FAVOR III China): a multicentre, randomised, sham-controlled trial. Lancet. 2021 Dec 11;398(10317):2149-2159. doi: 10.1016/S0140-6736(21)02248-0. Epub 2021 Nov 4. PMID 34742368
- [Background] Masdjedi K, van Zandvoort LJC, Balbi MM, Gijsen FJH, Ligthart JMR, Rutten MCM, Lemmert ME, Wilschut JM, Diletti R, de Jaegere P, Zijlstra F, Van Mieghem NM, Daemen J. Validation of a three-dimensional quantitative coronary angiography-based software to calculate fractional flow reserve: the FAST study. EuroIntervention. 2020 Sep 18;16(7):591-599. doi: 10.4244/EIJ-D-19-00466. PMID 31085504
- [Background] Fearon WF, Achenbach S, Engstrom T, Assali A, Shlofmitz R, Jeremias A, Fournier S, Kirtane AJ, Kornowski R, Greenberg G, Jubeh R, Kolansky DM, McAndrew T, Dressler O, Maehara A, Matsumura M, Leon MB, De Bruyne B; FAST-FFR Study Investigators. Accuracy of Fractional Flow Reserve Derived From Coronary Angiography. Circulation. 2019 Jan 22;139(4):477-484. doi: 10.1161/CIRCULATIONAHA.118.037350. PMID 30586699
- [Derived] Ki YJ, Hwang D, Yang S, Na SH, Doh JH, Nam CW, Kim DY, Choi BJ, Sohn CB, Lee HJ, Kim HK, Kim Y, Shin ES, Koo BK. Diagnostic Performance of Angiography-Derived FFR According to the Analysis Factors. Korean Circ J. 2025 Sep 3. doi: 10.4070/kcj.2025.0077. Online ahead of print. PMID 41044725